CLINICAL TRIAL: NCT00355030
Title: Efficacy and Safety of Somatropin in Combination With Leuprorelin Compared to Somatropin Alone in Pubertal Children With Idiopathic Short Stature
Brief Title: Somatropin + Leuprorelin vs Somatropin Alone in Pubertal Children With Idiopathic Short Stature
Acronym: Phoenix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9861; B9R-FP-GDGI (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Short Stature (ISS)
MeSH Terms: interventions — Human Growth Hormone; Growth Hormone; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: somatropin; Drug: leuprorelin
- 2 (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 0.05 mg/kg/day
  Other Names: LY137998; Humatrope
Drug: leuprorelin — 11.25 mg/3 months
  Arms: 1

SUMMARY:
The present randomized trial was initially intended to study the benefits of a combined treatment with growth hormone (GH) and a gonadotropin-releasing hormone (GnRH) agonist for pubertal children with idiopathic short stature. However, treatments were stopped in January 2012 at the request of the French drug agency. Therefore, a protocol amendment divided the study in two study periods.

Study Period 1 involved combined treatment with somatropin and leuprorelin or treatment with somatropin alone. Participants from France who participated in this Period 1 of the study were asked to participate in a long term safety follow up defined as a Period 2 of the study. Participants from the Netherlands were offered participation in Genetics and Neuroendocrinology of Short Stature International Study (GeNeSIS, clinicaltrials.gov Identifier: NCT01088412) for long term safety follow up independent of this study.

ELIGIBILITY:
Inclusion Criteria:

* male or female children with ISS
* age greater than or equal to 8 years and less than or equal to 12 years and 3 months for girls and greater than or equal to 9 years and less than or equal to 14 years and 3 months for boys
* bone age less than or equal to 12.0 years for girls and less than or equal to 14.0 years for boys based on a central reading of an X-ray of the left hand and wrist
* Pubertal stage B2 and B3 for girls based on the Tanner method
* Pubertal stage G2 and G3 for boys based on the Tanner method

Exclusion Criteria:

* Growth hormone deficiency (GHD)
* Insulin-like growth factor-I levels greater than 3 SDS
* Chromosomal abnormality diagnosed locally on a karyotype. For girls, the karyotype to eliminate a Turner syndrome, is mandatory
* Small for gestational age (SGA)
* Has reached menarche (had her first menstrual period)
* Have any significant concomitant disease that is likely to interfere with growth or with the study, or is a known contraindication to Growth Hormone treatment

Ages: 8 Years to 171 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2006-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- France (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boulogne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Havre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reims
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarbes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin and Leuprorelin: Experimental Arm 1: 0.05mg/kg/day subcutaneous somatropin and 3-month formulation, subcutaneous or intramuscular injection of 11.25mg leuprorelin for three years (or for a minimum of 2 years until a chronological age of 13 years for girls and 15 years for boys, whichever occurs first).
- Somatropin: Experimental Arm 2: 0.05mg/kg/day subcutaneous somatropin only
Period: Study Period 1 Treatment
Arm/Group | Somatropin and Leuprorelin: Experimental Arm 1 | Somatropin: Experimental Arm 2
Started | 46 | 45
Received At Least One Dose of Study Drug | 45 (1 non-eligible participant received somatropin from previous control group) | 43 (2 non-eligible participants received somatropin from previous control group)
Completed | 1 (Participants from the Netherlands exited the study after Study Period 1.) | 1 (Participants from the Netherlands exited the study after Study Period 1.)
Not Completed | 45 | 44
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Parent/Caregiver Decision | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Sponsor Decision | 34 | 32
Not completed — Protocol Entry Criterion Not Met | 0 | 1
Not completed — Other | 2 | 6
Period: Study Period 2 Long Term Follow-Up
Arm/Group | Somatropin and Leuprorelin: Experimental Arm 1 | Somatropin: Experimental Arm 2
Started | 20 (Participants from France were given the option to re-consent for Study Period 2.) | 19 (Participants from France were given the option to re-consent for Study Period 2.)
Completed | 19 | 17
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) includes all data from all randomized patients receiving at least one dose of the study drug according to the treatment to which the patients were assigned and with at least one follow-up visit.
Groups:
- Somatropin and Leuprorelin: 0.05mg/kg/day subcutaneous somatropin and 3-month formulation, subcutaneous or intramuscular injection of 11.25mg leuprorelin for three years (or for a minimum of 2 years until a chronological age of 13 years for girls and 15 years for boys, whichever occurs first).
- Somatropin: 0.05mg/kg/day subcutaneous somatropin only
- Total: Total of all reporting groups
Arm/Group | Somatropin and Leuprorelin | Somatropin | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (1.41) | 12.1 (1.33) | 12.1 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 19 | 23 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 6 | 5 | 11
  France | 39 | 38 | 77
Standing Height SDS [Mean (Standard Deviation); unit: Standard Deviation Score] | -2.5 (0.45) | -2.5 (0.46) | -2.5 (.045)
Standing Height [Mean (Standard Deviation); unit: centimeters] | 131.6 (6.72) | 131.6 (5.78) | 131.6 (6.24)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-related Adverse Events
Description: A drug-related AE was an AE that occurred postdose or was present predose and became more severe postdose and was considered to be related to study treatment. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through End of Study (up to 9 years)
Population: All participants who received at least one dose of study drug in Period 1 and all participants who entered Period 2 (safety population).
Measure: Number; unit: participants
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 46 | 45
participants
  Study Period 1 (n=46, 45) | 42 | 38
  Study Period 2 (n=20, 19) | 11 | 9

2. Primary Outcome: Adult Height Standard Deviation Score (SDS)
Description: The height of the participants were measured barefoot using a standard wall-mounted Harpenden stadiometer. SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End of Study (up to 9 years)
Population: All participants who received at least one dose of study drug with at least one follow up visit.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 19 | 16
standard deviation score | -1.8 (0.53) | -1.9 (0.77)

3. Secondary Outcome: Height Velocity
Description: Height velocity is the difference between 2 height measurements, divided by years elapsed between measurements.
Time Frame: Baseline through End of Study (up to 9 years)
Population: All participants who received at least one dose of study drug with at least one follow up visit. The safety follow up participants did not reach final height at end of Period 1 unless final height is noted for participants that reached final height at the end of Period 1.
Measure: Mean (Standard Deviation); unit: centimeter per year
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 45 | 43
centimeter per year
  Randomization (n=45, 43) | 7.8 (6.92) | 7.4 (6.03)
  Month 3 (n=45, 43) | 9.9 (3.94) | 10.6 (3.53)
  Month 6 (n=45, 42) | 8.1 (2.31) | 9.7 (2.80)
  Month 12 (n=44, 42) | 7.0 (1.64) | 8.8 (2.33)
  Month 18 (n=42, 42) | 6.6 (1.68) | 8.4 (2.64)
  Month 24 (n=37, 41) | 4.9 (1.33) | 7.8 (3.36)
  Month 30 (n=25, 25) | 6.2 (2.09) | 5.8 (2.93)
  Month 36 (n=18, 19) | 6.6 (3.25) | 3.5 (2.71)
  Month 42 (n=13, 14) | 5.7 (1.94) | 3.7 (2.17)
  Month 48 (n=7, 8) | 5.4 (2.27) | 2.9 (2.73)
  Month 54 (n=1, 1) | 6.3 (0) | 7.1 (0)
  Safety follow up 6 months (n=16, 9) | 4.6 (2.08) | 4.5 (2.45)
  Safety follow up 12 months(n=15, 8) | 2.9 (2.37) | 2.3 (1.43)
  Safety follow up 18 months (n=12, 4) | 3.3 (1.69) | 1.2 (1.20)
  Safety follow up 24 months (n=9, 1) | 2.0 (1.32) | 2.5 (0)
  Safety follow up 36 months (n=5, 0) | 1.3 (0.53) | 0 (0)
  Safety follow up 42 months (n=2, 0) | 2.1 (2.45) | 0 (0)
  Safety follow up 12 months (final height)(n=18,14) | 0.5 (0.86) | 0.8 (1.59)
  Safety follow up 24 months (final height) (n=7,10) | 0.3 (0.77) | 0.3 (0.97)
  Safety follow up 36 months (final height) (n=3,7) | 0.9 (0.78) | 0.3 (0.60)

4. Secondary Outcome: Height SDS
Description: SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End of Study (up to 9 years)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 45 | 43
standard deviation score
  Randomization (n=45, 43) | -2.5 (0.45) | -2.5 (0.46)
  Month 3 (n=45, 43) | -2.4 (0.42) | -2.4 (0.47)
  Month 6 (n=45, 42) | -2.3 (0.48) | -2.2 (0.52)
  Month 12 (n=44, 42) | -2.2 (0.50) | -2.0 (0.57)
  Month 18 (n=42, 42) | -2.2 (0.53) | -1.9 (0.63)
  Month 24 (n=37, 41) | -2.3 (0.58) | -1.8 (0.67)
  Month 30 (n=25, 25) | -2.2 (0.63) | -2.0 (0.58)
  Month 36 (n=18, 19) | -2.0 (0.65) | -2.0 (0.68)
  Month 42 (n=13, 14) | -1.8 (0.68) | -1.9 (0.66)
  Month 48 (n=7, 8) | -1.6 (0.52) | -1.9 (0.65)
  Month 54 (n=1, 1) | -1.0 (0) | -1.7 (0)
  Safety follow up 6 months (n=16, 9) | -2.1 (0.65) | -1.7 (0.77)
  Safety follow up 12 months(n=15, 8) | -1.9 (0.55) | -1.7 (0.77)
  Safety follow up 18 months (n=12, 4) | -1.9 (0.63) | -1.9 (0.78)
  Safety follow up 24 months (n=9, 1) | -1.9 (0.46) | -1.2 (0)
  Safety follow up 36 months (n=5, 0) | -1.9 (0.67) | 0 (0)
  Safety follow up 42 months (n=2, 0) | -2.4 (0.18) | 0 (0)
  Safety follow up 12 months (final height)(n=18,14) | -1.9 (0.46) | -1.8 (0.71)
  Safety follow up 24 months (final height) (n=7,10) | -1.6 (0.56) | -2.0 (0.79)
  Safety follow up 36 months (final height) (n=3,7) | -1.2 (0.90) | -2.2 (0.94)

5. Secondary Outcome: Difference Between Adult Height SDS and Target Height SDS
Description: This is the difference between the gender, age and country matched standard deviation score of adult height and standard deviation score of target height [calculated as (mother's height (SDS) + father's height (SDS))/2] for particular participant.
  The height of the participants were measured barefoot using a standard wall-mounted Harpenden stadiometer. SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End of Study (up to 9 years)
Population: All participants who received who reached final height.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 16 | 15
standard deviation score | -0.6 (0.89) | -1.2 (0.80)

6. Secondary Outcome: Difference Between Adult Height SDS and Baseline Predicted Height SDS
Description: This is the difference between the gender, age and country matched standard deviation score of adult height and standard deviation score of baseline predicted height [calculated using the Bayley-Pinneau method based on height and bone age] for particular participant.
  The height of the participants were measured barefoot using a standard wall-mounted Harpenden stadiometer. SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End up Study (up to 9 years)
Population: All participants who received who reached final height.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 18 | 16
standard deviation score | 1.1 (0.96) | 1.2 (0.70)

7. Secondary Outcome: Difference Between Adult Height SDS and Baseline Height SDS
Description: This is the difference between the gender, age and country matched standard deviation score of adult height and standard deviation score of baseline height for particular participant.
  The height of the participants were measured barefoot using a standard wall-mounted Harpenden stadiometer. SDS report the number of standard deviations from the mean for age and sex for an individual measurement (normal range: -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End up Study (up to 9 years)
Population: All participants who received who reached final height.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 19 | 16
standard deviation score | 0.6 (0.59) | 0.6 (0.67)

8. Secondary Outcome: Percentage of Children With Normal Adult Height SDS
Description: Percentage of children with normal adult height SDS (greater than -2 SDS and less than +2 SDS)
Time Frame: Baseline through End of Study (up to 9 years)
Population: All participants who received at least one dose of study drug with at least one follow up visit.
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 45 | 43
percentage of participants | 26.7 | 25.6

9. Secondary Outcome: Bone Age
Description: Bone age measured using the X-Ray of left hand and wrist.
Time Frame: Baseline through End of Study (up to 9 years)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Somatropin and Leuprorelin | Somatropin
Number analyzed (Participants) | 45 | 43
years
  Randomization (n=45, 43) | 10.8 (1.58) | 11.0 (1.45)
  Month 12 (n=40, 41) | 11.7 (1.59) | 12.1 (1.12)
  Month 24 (n=34, 37) | 12.4 (1.32) | 13.4 (1.09)
  Month 36 (n=18, 18) | 13.3 (1.49) | 14.5 (1.64)
  Month 48 (n=7, 8) | 14.8 (1.33) | 15.4 (1.27)
  Safety follow up 6 months (n=16, 7) | 14.1 (1.11) | 14.9 (0.81)
  Safety follow up 18 months (n=12, 3) | 15.2 (1.25) | 17.0 (1.00)
  Safety follow up 36 months (n=5, 0) | 15.7 (1.04) | 0 (0)
  Safety follow up 12 months (final height)(n=18,14) | 19.6 (14.53) | 16.3 (1.27)

ADVERSE EVENTS:
Groups:
- Somatropin and Leuprorelin: Somatropin and leuprorelin n=46
- Somatropin: Somatropin n=45
Arm/Group | Somatropin and Leuprorelin | Somatropin
Serious Adverse Events (participants affected / at risk) | 12/46 | 7/45
Other Adverse Events (participants affected / at risk) | 41/46 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin and Leuprorelin (N=46) | Somatropin (N=45)
Congenital genital malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin and Leuprorelin (N=46) | Somatropin (N=45)
Ear pain (Ear and labyrinth disorders) | 1 (5) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (18)
Abdominal pain upper (Gastrointestinal disorders) | 3 (11) | 4 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (14) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (7) | 2 (3)
Toothache (Gastrointestinal disorders) | 3 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (5)
Injection site pain (General disorders) | 8 (22) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 5 (6)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 4 (4) | 5 (8)
Gastroenteritis (Infections and infestations) | 11 (15) | 6 (9)
Influenza (Infections and infestations) | 15 (17) | 9 (16)
Nasopharyngitis (Infections and infestations) | 19 (36) | 8 (10)
Rhinitis (Infections and infestations) | 5 (5) | 3 (11)
Tonsillitis (Infections and infestations) | 6 (9) | 5 (12)
Tracheitis (Infections and infestations) | 2 (2) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 21 (51) | 16 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (6)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (7)

LIMITATIONS AND CAVEATS:
No statistical analyses was performed after the early treatment termination. All data represented is descriptive statistics only and no confirmatory conclusions can be drawn from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days